CLINICAL TRIAL: NCT00035347
Title: A Randomized, Multicenter, Open Label Trial Comparing Intravenous Zithromax® (Azithromycin) Plus Intravenous Rocephin® (Ceftriaxone) Followed By Oral Zithromax® (Azithromycin) With Intravenous Levaquin® (Levofloxacin) Followed By Oral Levaquin® (Levofloxacin) For The Treatment Of Moderate To Severely Ill Hospitalized Subjects With Community-Acquired Pneumonia
Brief Title: Intravenous Azithromycin Plus Intravenous Ceftriaxone Followed by Oral Azithromycin With Intravenous Levofloxacin Followed by Oral Levofloxacin for the Treatment of Moderate to Severely Ill Hospitalized Patients With Community Acquired Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661035
Record Dates: First submitted 2002-05-02; First posted 2002-05-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Community-Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Azithromycin; Ceftriaxone; Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azithromycin plus ceftriaxone group (AZY+CEF group) (Experimental): IV azithromycin (500 mg once daily) plus ceftriaxone (1 gram once daily) for 2 to 5 days followed by oral azithromycin (2 x 250 mg once daily) to complete a total of 7 to 10 days of therapy
  Interventions: Drug: IV azithromycin; Drug: ceftriaxone; Drug: oral azithromycin
- Levofloxacin group (LEV group) (Experimental): IV levofloxacin (500 mg once daily) for a minimum of 2 days followed by oral levofloxacin (500 mg once daily) to complete a total of 7 to 14 days of therapy.
  Interventions: Drug: IV levofloxacin; Drug: oral levofloxacin

INTERVENTIONS:
Drug: IV azithromycin — 500 mg once daily
  Other Names: Zithromax®
  Arms: Azithromycin plus ceftriaxone group (AZY+CEF group)
Drug: ceftriaxone — 1 gram once daily for 2 to 5 days
  Other Names: Rocephin®
  Arms: Azithromycin plus ceftriaxone group (AZY+CEF group)
Drug: oral azithromycin — 2 x 250 mg once daily
  Other Names: Zithromax®
  Arms: Azithromycin plus ceftriaxone group (AZY+CEF group)
Drug: IV levofloxacin — 500 mg once daily
  Other Names: Levaquin®
  Arms: Levofloxacin group (LEV group)
Drug: oral levofloxacin — 500 mg once daily
  Other Names: Levaquin®
  Arms: Levofloxacin group (LEV group)

SUMMARY:
A trial in which patients over 18 years of age who are hospitalized with community acquired pneumonia and are otherwise eligible for entry into the study are randomly selected to receive one of two treatment regimens. After written informed consent is obtained, patients will receive one of the following two treatment regimens: 1) intravenous administration of azithromycin and ceftriaxone followed by azithromycin tablets, or 2) intravenous administration of levofloxacin followed by levofloxacin tablets. At least four study visits are normally conducted up to approximately one month after starting therapy. The objective of this study is to compare the safety and efficacy of the two treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older.
* Patient must be hospitalized and require intravenous therapy for treatment of pneumonia.
* Patient must have pneumonia as documented by relevant signs and symptoms and a positive chest X-ray.
* Patients cannot have certain underlying diseases or conditions as defined in the study protocol.

Exclusion Criteria:

* Pregnant women, nursing mothers, or women of childbearing potential not practicing adequate contraception.
* Known or suspected hypersensitivity or intolerance to any quinolone, penicillin, cephalosporin, or macrolide antibiotic.
* Treatment with any systemic antibiotic for 24 hours or longer within 72 hours prior to the baseline visit.
* Subjects with clinically significant renal dysfunction.
* Subjects with clinically significant hepatic dysfunction.
* Subjects with clinically significant cardiovascular disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2001-01; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of sequential therapy with IV Zithromax® plus IV Rocephin® followed by oral Zithromax® to IV Levaquin® (levofloxacin) followed by oral Levaquin® in the treatment of moderate to severely ill subjects with community-acquired pneumonia. | Duration of trial

SECONDARY OUTCOMES:
Safety and toleration of IV Zithromax® plus IV Rocephin® followed by oral Zithromax® to IV Levaquin® followed by oral Levaquin®, and to compare the bacteriological response rates in subjects with a baseline pathogen. | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (21):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Sylmar, California
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Fort Eisenhower, Georgia
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Kirkwood, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, San Antonio, Texas
- Canada (9):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Germany (3):
  - Pfizer Investigational Site, Rotenburg (Wümme), Lower Saxony
  - Pfizer Investigational Site, Berlin, State of Berlin
  - Pfizer Investigational Site, Lüdenscheid
- Pfizer Investigational Site, Maroussi. Attikis, Athens, Greece
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Catalonia
  - Pfizer Investigational Site, Tarrasa, Catalonia